CLINICAL TRIAL: NCT06094699
Title: Improving Sleep in the Neurology In-Patient Population
Acronym: I_SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Laura Stein, Principal Investgiator, University of Pennsylvania
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 850574
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention)
- Sleep intervention (Experimental)
  Interventions: Other: Sleep friendly order set; Other: Patient sleep menu

INTERVENTIONS:
Other: Sleep friendly order set — Every evening, the following orders (which comprise the sleep-friendly order set) will be input into the EMR:
  Hold vital signs and neurological checks overnight Retime applicable medications outside of the nighttime window of 10pm-6am Retime daily lab draws outside of the nighttime window of 10pm-6am Order melatonin if no clinical contraindications Discontinue finger stick glucose measurements for patients with a stable blood glucose values Change DVT prophylaxis to enoxaparin for all clinically eligible patients
  Arms: Sleep intervention
Other: Patient sleep menu — Patients will be given a menu of non-pharmacological options that support sleep by improving comfort and reducing anxiety.
  Arms: Sleep intervention

SUMMARY:
We aim to test multiple interventions to improve sleep for Neurology inpatients, including 1) a sleep-friendly order set, and 2) a sleep menu. We will collect patient sleep data, including duration and quality, via actigraphy devices (FitBits). We will also conduct qualitative patient surveys to understand the impact of these interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* 24 hours after admission to the general neurology (ward) service at the Hospital of the University of Pennsylvania
* Patients who are determined by the primary team to be clinically stable enough to forego serial overnight vital signs monitoring and neuro checks.
* Clinical stability criteria:
* Symptomatic stability >24h after admission (no new or progressive neurologic symptoms for >24 hours)
* Vital signs stability on admission for > 24h while admitted
* Ability to verbally consent to study participation

Exclusion Criteria:

* Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Any additional clinical factors felt by the team to be incompatible with specific orders including requiring serial vital signs monitoring and neuro checks overnight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Fitbit Sleep Duration | Duration of hospitalization from consent to discharge or day 10, whichever comes first
  Total hours of sleep

SECONDARY OUTCOMES:
FitBit sleep score | Duration of hospitalization from consent to discharge or day 10, whichever comes first
  The sleep score integrates subject sleep deprivation, sleep depth, and sleep restoration
Richard Campbell Sleep Questionnaire (RCSQ) | Duration of hospitalization from consent to discharge or day 10, whichever comes first
  The Richards-Campbell Sleep Questionnaire (RCSQ) is a simple, validated survey instrument for measuring sleep quality in intensive care patients
Patient reported Sleep Duration and Quality | Duration of hospitalization from consent to discharge or day 10, whichever comes first
  A brief survey collecting patient perceived duration and quality of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Laura Stein, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States